CLINICAL TRIAL: NCT01082705
Title: Impact Tanzania in Vivo Efficacy 2010: Assessing the Efficacy of Artemisinin Combination Therapies for Treatment of Uncomplicated Malaria Infection in Children Aged 6-59 Months
Brief Title: Assessing the Efficacy of Artemisinin Combination Therapies for Treatment of Uncomplicated Malaria Infection in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Julie Gutman, Medical Epidemiologist, Malaria Branch, Centers for Disease Control and Prevention
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMPACT TZ IV2010
Record Dates: First submitted 2010-03-08; First posted 2010-03-09 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: P. Falciparum Malaria
Keywords: malaria; treatment; artemisinin combination therapy; Tanzania; P. falciparum malaria in children age 6-59 months
MeSH Terms: conditions — Malaria | interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Artemether-lumefantrine (Active Comparator): Artemether-lumefantrine (Coartem; Novartis) administered twice daily for three days as tablets containing 20 mg of artemether plus 120 mg of lumefantrine at a dosage of: 1 tablet for patients weighing 5-14 kg, 2 tablets for patients weighing 15-24 kg, 3 tablets for patients weighing 25-34 kg, 4 tablets for patients weighing 35 kg or more
  Interventions: Drug: artemether-lumefantrine
- Dihydroartemisinin-piperaquine (Experimental): Dihydroartemisinin-piperaquine administered once daily for 3 days as tablets containing 40 mg of dihydroartemisinin and 320 mg of piperaquine at a total dosage of 6.4 mg/kg of dihydroartemisinin and 51.2 mg/kg of piperaquine divided equally between the three days
  Interventions: Drug: Dihydroartemisinin-piperaquine

INTERVENTIONS:
Drug: artemether-lumefantrine — administered twice daily for three days as tablets containing 20 mg of artemether plus 120 mg of lumefantrine at a dosage of: 1 tablet for patients weighing 5-14 kg, 2 tablets for patients weighing 15-24 kg, 3 tablets for patients weighing 25-34 kg, 4 tablets for patients weighing 35 kg or more
  Other Names: Coartem Novartis
  Arms: Artemether-lumefantrine
Drug: Dihydroartemisinin-piperaquine — once daily for 3 days as tablets containing 40 mg of dihydroartemisinin and 320 mg of piperaquine at a total dosage of 6.4 mg/kg of dihydroartemisinin and 51.2 mg/kg of piperaquine divided equally between the three days
  Arms: Dihydroartemisinin-piperaquine

SUMMARY:
Following the rapid development of significant drug resistance to both chloroquine and sulfadoxine-pyrimethamine (the first line therapy in Tanzania from 2001 -2006), artemether- lumefantrine (Coartem or AL) was adopted as first line therapy in Tanzania in 2006. Now that this drug has been widely used for some time, the investigators propose to conduct an antimalarial efficacy trial to monitor the effectiveness of this therapy, to determine if this drug remains efficacious, or if significant resistance has emerged, in which case a new antimalarial strategy will need to be contemplated. The investigators hypothesize that the efficacy of Artemether-lumefantrine remains high, and that the other artemisinin combination therapies will be equally efficacious.

Children 6-59 months of age with symptomatic malaria will be randomly assigned to be treated with either artemether + lumefantrine (Coartem) or dihydroartemisinin-piperaquine (Duo-Cotecxin or Artekin). Clinical, parasitologic, and hematologic parameters will be monitored over a 42-day follow-up period and will be used to evaluate drug efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 6-59 months
2. Axillary temperature ≥ 37.5º C or history of fever in the past 48 hours
3. Weight ≥ 5.0 kg
4. Slide-confirmed infection with P. falciparum, with parasitemia 2,000-200,000 asexual forms per μl
5. Live within the boundaries of the officially recognized catchment area of Miono Health Center.
6. Caregiver agrees to all blood draws and return visits.

Exclusion Criteria:

1. General danger signs or symptoms of severe malaria
2. Signs or symptoms of severe malnutrition, defined as weight-for-age ≤ 3 standard deviations below the mean (National Center for Health Statistics [NCHS]/World Health Organization [WHO] normalized reference values)
3. Slide confirmed infection with any other Plasmodium spp. besides falciparum or mixed plasmodium infection
4. Severe anemia, defined as Hb < 5 g/dl
5. Known hypersensitivity to any of the drugs being tested
6. Presence of febrile conditions caused by diseases other than malaria
7. Serious or chronic medical condition (heart failure, sickle cell disease).
8. Plan to travel or leave the area within the next 3 months.
9. Have been treated for malaria in the 2 weeks prior to enrollment.

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 323 (Actual)
Dates: Start 2010-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
42-day polymerase chain reaction (PCR)-adjusted parasitological cure of P. falciparum parasitemia | 42 days

SECONDARY OUTCOMES:
Hematologic response to treatment measured as mean change in hemoglobin concentration from Day 0 to Day 42 | 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Julie R Gutman, MD MSc, Study Director — Centers for Disease Control and Prevention; S. Patrick Kachur, MD MPH, Principal Investigator — Centers for Disease Control and Prevention
Locations (1):
- Miono Health Center, Bagamoyo, Tanzania